CLINICAL TRIAL: NCT01516437
Title: A Study to Assess Immunity to Specific Microbial Antigens in Healthy Smokers and Non-smokers and in Subjects With Stable Chronic Obstructive Pulmonary Disease (COPD) Aged Between 45-75 Years
Brief Title: A Study to Assess Immunity to Specific Microbial Antigens in Healthy Smokers and Non-smokers and in Subjects With Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 116021
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Disorders
Keywords: Chronic Obstructive Pulmonary disease (COPD)
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection

ARMS (4):
- HNS Group (Experimental): Healthy non-smokers aged between 45-75 years
  Interventions: Procedure: Blood collection; Procedure: Swab collection
- HS Group (Experimental): Healthy smokers aged between 45-75 years
  Interventions: Procedure: Blood collection; Procedure: Swab collection
- FeCOPD Group (Experimental): COPD subjects with ≥ two exacerbations within 365 days prior to the screening visit (frequent exacerbators), aged between 45-75 years
  Interventions: Procedure: Blood collection; Procedure: Swab collection; Procedure: Sputum collection
- NFeCOPD Group (Experimental): COPD patients with one exacerbation within 365 days prior to the screening visit (non-frequent exacerbators), aged between 45-75 years
  Interventions: Procedure: Blood collection; Procedure: Swab collection; Procedure: Sputum collection

INTERVENTIONS:
Procedure: Blood collection — Blood collection at Day 0 (all subjects) and at Month 6 (COPD subjects) for the analysis of serology, cell-mediated immune response.
Procedure: Swab collection — Nasopharyngeal and oropharyngeal swabs collection at Day 0 (All subjects) and at exacerbation visits (COPD subjects).
Procedure: Sputum collection — Sputum collection at Day 0 and at exacerbation visits (COPD subjects)
  Arms: FeCOPD Group; NFeCOPD Group

SUMMARY:
The present study aims to assess the natural immunity to specific microbial antigens in healthy subjects and in subjects with stable COPD aged between 45-75 years.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects (smokers and non-smokers)

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including 45 and 75 years of age at the time of consent.
* Written informed consent obtained from the subject.
* Baseline post-bronchodilator Forced Expiratory Volume of air in one second (FEV1) > 85% of predicted normal values and baseline post-bronchodilator FEV1/Forced expiratory Vital Capacity (FVC) > 70% of predicted normal values.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Non-smokers: subjects who never smoked OR
* Smokers: current smoker having a smoking history ≥ 10 pack-years.

COPD subjects (frequent and non-frequent exacerbators)

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including 45 and 75 years of age at the time of consent.
* Written informed consent obtained from the subject.
* Baseline post-bronchodilator FEV1 < 80% and >30% of predicted normal values and baseline post-bronchodilator FEV1/FVC < 70% of predicted normal values.
* Current or former smoker having a smoking history of ≥ 10 pack-years.
* Documented history of ≥ one exacerbation within 365 days prior to the screening visit that required treatment with systemic corticosteroids or resulted in hospitalization.

Exclusion Criteria:

Healthy subjects (smokers and non-smokers)

* Use of any investigational or non-registered product within 30 days prior to Screening Visit or planned use during the study.
* Concurrently participating in another clinical study in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any known clinically significant anaemia or any other condition as per medical records that would preclude the drawing of blood as described in the protocol.
* Receipt of any vaccine within 30 days preceding blood sampling.
* Previous vaccination with any NTHi vaccine.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 180 days prior to screening visit. Topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Any known respiratory disorders.
* Acute disease and/or fever at the time of the Screening Visit or Visit 1, as applicable
* Receipt of immunoglobulins and/or any blood products within 90 days prior to Screening Visit.
* Receipt of interferon within 90 days prior to Screening Visit.
* History of malignancy.
* Subjects with a history of, or current, alcohol or substance abuse.
* Known history of immune-mediated disorder.
* Recent use of antibiotics or antiviral drug within 30 days prior to Screening Visit.
* Pregnant female.
* Other conditions that the investigator judges may interfere with study findings.

COPD subjects (frequent and non-frequent exacerbators)

* Use of any investigational or non-registered product within 30 days prior to Screening Visit or planned use during the study. Use of investigational inhaled long acting muscarinic antagonists (LAMA), inhaled long acting beta agonists (LABA) or inhaled corticosteroids is allowed.
* Concurrently participating in another clinical study in which the subject has been or will be exposed to an investigational or a non-investigational product. Subjects participating in clinical studies with investigational inhaled LAMA and/or LABA and/or inhaled corticosteroids can be enrolled.
* Any known clinically significant anaemia or any other condition as per medical records that would preclude the drawing of blood as described in the protocol.
* Receipt of any vaccine within 30 days preceding blood sampling.
* Previous vaccination with any NTHi vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* Serious, uncontrolled disease likely to interfere with the study findings.
* Acute disease and/or fever at the time of the Screening Visit or Visit 1, as applicable
* Receipt of immunoglobulins and/or any blood products within 90 days prior to Screening Visit.
* Receipt of interferon within 90 days prior to Screening Visit.
* History of malignancy.
* Subjects with a history of, or current, alcohol or substance abuse.
* Known history of immune-mediated disease other than COPD.
* Recent use of antibiotics or antiviral drug within 30 days prior to Screening Visit.
* Subject who experienced COPD exacerbation which required antibiotic, systemic corticosteroid or hospitalisation and which did not resolve at least one month prior to Screening Visit and at least 30 days following the last dose of oral corticosteroids.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 180 days preceding screening visit.
* Subjects with very severe COPD, GOLD stage IV.
* Primary diagnosis of asthma.
* Other respiratory disorders such as sarcoidosis, tuberculosis, lung cancer, lung fibrosis, cystic fibrosis.
* A known diagnosis of α-1 antitrypsin deficiency as underlying cause of COPD.
* History of lung surgery.
* Pregnant female.
* Other conditions that the investigator judges may interfere with study findings.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-06-28 (Actual); Study Completion 2012-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms. 3 enrolled subjects did not receive subject allocations, and were excluded from the study prior to start.
Period: Overall Study
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Started | 24 | 24 | 15 | 7
Completed | 24 | 24 | 14 | 6
Not Completed | 0 | 0 | 1 | 1
Not completed — Reason not specified | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group | Total
Number analyzed (Participants) | 24 | 24 | 15 | 7 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (10.10) | 57.8 (8.45) | 64.1 (7.39) | 61.4 (6.75) | 60.26 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 6 | 2 | 33
  Male | 8 | 15 | 9 | 5 | 37

OUTCOME MEASURES:

1. Primary Outcome: Anti-protein D Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per millilitre (EU/mL)
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol cohort at Day 0, which included all evaluable subjects for whom at least one assay results was available for the blood samples collected at Day 0.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 23 | 24 | 15 | 7
EU/mL | 79.5 [50.2 to 126.0] | 66.9 [53.1 to 84.3] | 61.7 [48.3 to 78.7] | 72.8 [40.1 to 132.0]

2. Primary Outcome: Anti-protein D Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL)
Time Frame: At Month 6
Population: The analysis was performed on the According-to-Protocol cohort at Month 6, which included all evaluable subjects for whom at least one assay results was available for the blood samples collected at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 13 | 6
EU/mL | 68.6 [50.2 to 93.9] | 61.0 [36.6 to 101.8]

3. Primary Outcome: Anti-Pneumococcal Histidine Triad D Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
EU/mL | 3786.7 [2748.3 to 5217.5] | 3400.7 [2445.3 to 4729.4] | 3323.9 [2128.8 to 5190.1] | 2563.9 [840.5 to 7821.6]

4. Primary Outcome: Anti-Pneumococcal Histidine Triad D Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL)
Time Frame: At Month 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 14 | 6
EU/mL | 2521.5 [1598.6 to 3977.4] | 2160.1 [863.2 to 5405.5]

5. Primary Outcome: Anti-pneumolysin Antibody Concentrations
Description: The analysis was performed on the According-to-Protocol cohort at Day 0, which included all evaluable subjects for whom at least one assay results was available for the blood samples collected at Day 0.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
EU/mL | 3870.5 [2607.0 to 5746.3] | 3116.7 [2097.3 to 4631.8] | 2804.5 [1831.8 to 4293.7] | 3898.7 [1437.4 to 10574.5]

6. Primary Outcome: Anti-pneumolysin Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EU/mL)
Time Frame: At Month 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 14 | 6
EU/mL | 2275.6 [1344.0 to 3853.0] | 3222.3 [1416.5 to 7330.4]

7. Primary Outcome: Concentrations for Serum Protein-D Enzymatic Inhibition
Description: Concentrations are presented as geometric mean concentrations (GMCs). The reference seropositivity cut-off value was ≥ 17.8%.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
EU/mL | 10.4 [8.9 to 12.1] | 9.3 [8.5 to 10.0] | 9.9 [8.4 to 11.7] | 8.9 [8.9 to 8.9]

8. Primary Outcome: Concentrations for Serum Protein-D Enzymatic Inhibition
Description: as for outcome 7
Time Frame: At Month 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 14 | 6
EU/mL | 9.4 [8.4 to 10.4] | 8.9 [8.9 to 8.9]

9. Primary Outcome: Number of Subjects With PD Enzymatic Inhibition Concentration Greater Than or Equal to (≥) 17.8%
Description: Concentrations were expressed as geometric mean concentrations (GMCs)
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
Subjects | 4 | 1 | 2 | 0

10. Primary Outcome: Number of Subjects With PD Enzymatic Inhibition Concentration Greater Than or Equal to (≥) 17.8%
Description: Concentrations were expressed as geometric mean concentrations (GMCs)
Time Frame: At Month 6
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 14 | 6
Subjects | 1 | 0

11. Secondary Outcome: Frequency of Specific Cluster of Differentiation 4+ (CD4+) T Cells Expressing at Least 2 Markers Among CD 40 Ligand (CD40L), Interleukin 2 (IL-2), Tumor Necrosis Factor-α (TNF-α), Interferon-γ (IFN-γ), IL-13 and IL-17 Upon in Vitro Stimulation
Time Frame: At Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
T cells/million cells | 159.6 (67.29) | 163.5 (87.11) | 173.9 (89.69) | 170.1 (88.96)

12. Secondary Outcome: Frequency of Specific Cluster of Differentiation 8+ (CD8+) T Cells Expressing at Least 2 Markers Among CD 40 Ligand (CD40L), Interleukin 2 (IL-2), Tumor Necrosis Factor-α (TNF-α), Interferon-γ (IFN-γ), IL-13 and IL-17 Upon in Vitro Stimulation
Time Frame: At Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
T cells/million cells | 97.9 (56.74) | 125.2 (73.93) | 125.2 (44.12) | 161.3 (43.72)

13. Secondary Outcome: Number of Subjects With Positive Sputum - Culture Testing Results
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 15 | 7
Subjects
  Any bacteria | 9 | 1
  Streptococcus pneumoniae | 0 | 0
  Haemophilus influenzae | 2 | 1
  Moraxella catarrhalis | 2 | 0
  Staphylococcus aureus | 1 | 0
  Pseudomonas aeruginosa | 0 | 0
  Other bacteria | 6 | 0

14. Secondary Outcome: Number of Subjects With Positive Nasopharyngeal Swab - Culture Testing Results
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
Subjects
  Any bacteria | 4 | 1 | 4 | 0
  Streptococcus pneumoniae | 0 | 1 | 0 | 0
  Haemophilus influenzae | 0 | 0 | 0 | 0
  Moxarella catarrhalis | 0 | 0 | 0 | 0
  Staphylococcus aureus | 4 | 0 | 3 | 0
  Pseudomonas aeruginosa | 0 | 0 | 0 | 0
  Other bacteria | 0 | 0 | 1 | 0

15. Secondary Outcome: Number of Subjects With Positive Oropharyngeal Swab - Culture Testing Results
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Number analyzed (Participants) | 24 | 24 | 15 | 7
Subjects
  Any bacteria | 5 | 3 | 5 | 1
  Streptococcus pneumoniae | 0 | 1 | 0 | 0
  Haemophilus influenzae | 2 | 1 | 2 | 0
  Moxarella catarrhalis | 0 | 0 | 0 | 0
  Staphylococcus aureus | 1 | 1 | 1 | 0
  Pseudomonas aeruginosa | 0 | 0 | 0 | 0
  Other bacteria | 2 | 0 | 4 | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) up to Month 6.
Description: Non-serious/frequent adverse events were not collected in this study.
Arm/Group | HNS Group | HS Group | FeCOPD Group | NFeCOPD Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 1/15 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HNS Group (N=24) | HS Group (N=24) | FeCOPD Group (N=15) | NFeCOPD Group (N=7)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.